CLINICAL TRIAL: NCT04290611
Title: Monitoring the Neurological Toxicity of Enzalumatide Through VigiBase, a Pharmacovigilance Study
Brief Title: a Vigibase Pharmacovigilance Study of ENzalutamide Drug-induced neurotoxicitY
Acronym: VENDY
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Principal Investigator, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-20-02
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer; Neuropathy; Epilepsy; Encephalopathy
Keywords: Drug-induced neurotoxicity
MeSH Terms: conditions — Prostatic Neoplasms; Epilepsy; Brain Diseases | interventions — enzalutamide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Enzalutamide drug-induced toxicity: Cases reported in the World Health Organization (WHO) and the French pharmacovigilance database of patients treated by enzalutamide, with a chronology compatible with the drug toxicity
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide for the treatment of prostate cancer or other solid tumors

SUMMARY:
Enzalutamide may lead to various adverse reactions. This study investigates reports of different neurological toxicities in the World Health Organization's (WHO) global database of individual safety case reports (VigiBase).

DETAILED DESCRIPTION:
Enzalutamide are responsible of a wide range of side effects.The investigators use VigiBase, the World Health Organization (WHO) database of individual safety case reports, to identify cases of adverse drug reactions following treatment with enzalutamide

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/01/2020 Adverse events reported were including any MedDRA terms Patients treated with enzalutamide reported in the WHO database.

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with enzalutamide for prostate cancer or other solid tumors
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with neurological adverse events with significant over-reporting enzalutamide | Case reported in the World Health Organization (WHO) of individual safety case reports to January 2020
  Identification and report of neurological toxiciy of enzalutamdie

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigation Clinique Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No